CLINICAL TRIAL: NCT03156686
Title: SAFEty and Efficacy of HOME-based Hospitalization Versus Inpatient Care for Patients With Acute Heart Failure in Chronic Heart Failure.
Acronym: SAFE-HOME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator couldn't include enough patients
Sponsor: French Cardiology Society (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-07
Record Dates: First submitted 2017-04-24; First posted 2017-05-17 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
Keywords: Acute Heart Failure; Chronic Heart Failure; Home care services; Cost-Benefit Analysis; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will be randomly assigned to conventional hospital care
- Home care treatment (Experimental): Patients will be randomly assigned to the HOME-based hospitalization and treated with intravenous diuretics. Following discharge within 48 hours from the hospital, patients in the HC group will be treated at home.
  Interventions: Procedure: HOME-based hospitalization

INTERVENTIONS:
Procedure: HOME-based hospitalization — patients in Home care treatment (HC) group will be treated at home
  Arms: Home care treatment

SUMMARY:
Evaluation of the efficacy, safety and and cost of home care versus conventional hospitalization care at 3-months in patients with worsening chronic heart failure.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) has an important socio-economic impact due to frequent hospital readmissions.

Hypothesis: Home care treatment (HC) will improve quality of live and decrease cost.

Methodology: Pilot, prospective, open, randomized controlled trial with 1-year follow-up for CHF patients admitted to 10 French hospital from March 2017 through February 2018, for acute decompensation of CHF. Patients will be randomly assigned to conventional hospital care or to the HC and treated with intravenous diuretics. Following discharge within 48 hours from the hospital, patients in the HC group will be treated at home. Follow-up will be conducted for both groups at discharge, 3 and 12 months after inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure (with history of Chronic Heart Failure)
* Identified in the first 48 hours
* Eligible for home-care with "Hospitalisation à Domicile" within 4 days after hospitalization.
* Patient affiliated to social security and to complementary health insurance

Exclusion Criteria:

* Under 18 years old
* Predominantly left-sided heart failure, dependent on oxygen because of the congestion
* Unexplored heart failure, indication of specific techniques (angiography) of device implantations (ICD, CRT).
* Severe cognitive disorders. Behavior disorders.
* Severe renal dysfunction with eGFR (MDRD) < 15 mL/min/1.73m2
* Patient leaving alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time to rehospitalization | within the first 3 months after the randomization.
  Time to rehospitalization for a new episode of acute heart failure within the first 3 months after the randomization.

SECONDARY OUTCOMES:
Occurrence of adverse events | during hospitalization at the end of the IV treatment which will be different for each patient, average of 15 days
  Occurrence of adverse events evaluated at the end of the IV treatment which will be different for each patient.
Quality of life (scales) | at the end of the treatment and 3 months
  Quality of life (scales) at the end of the treatment and 3 months
Nutritional status | at the end of the treatment and 3 months
  Evaluation of the nutritional status based on MNA score at the beginning of the IV treatment and 3 months and dietary survey at the beginning and the end of the IV treatment.
Mortality at the end of the treatment, 3 months and 1 year | at the end of the treatment, 3 months and 1 year
  Mortality at the end of the treatment, 3 months and 1 year
Cost-effectiveness | at the end of the treatment, 3 months and 1 year
  Cost-effectiveness at the end of the treatment, 3 months and 1 year
Time to first rehospitalization | within the first year after the randomization.
  Time to first rehospitalization for a new episode of acute heart failure within the first year after the randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud DAMY, MD, Principal Investigator — CH HENRI MONDOR
Locations (2):
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No